CLINICAL TRIAL: NCT01441466
Title: Cross-infection in Children Hospitalized for Bronchiolitis: Incidence, Symptoms en Effect of Cohort Isolation
Brief Title: Cohort Isolation and Cross-infection in Bronchiolitis
Status: Completed | Type: Observational
Sponsor: Princess Amalia Children's Clinic (Other)
Responsible Party: Principal Investigator, Jolita Bekhof, MD, Pediatrician, Princess Amalia Children's Clinic
Other Study IDs: bronchiolitis
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-01

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; RSV
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group without isolation: Patients in this arm are nursed together (in the same room) independent of viral agent.
  Interventions: Other: Isolation
- group with isolation: Patients in this arm are nursed separately until the test result of the PCR (polymerase chain reaction) for viral agents is known (within 24-48 hrs). RS-positive patients are nursed separately (separate room) from RS-negative patients

INTERVENTIONS:
Other: Isolation — Patients in this arm are nursed together (in the same room) independent of viral agent
  Groups: Group without isolation

SUMMARY:
The purpose of this study is to investigate the effect of cohort isolation of RS(respiratory syncytial virus)-positive bronchiolitis versus RS-negative bronchiolitis on prevention of co-infection and clinical disease severity. Furthermore the investigators want to elucidate general epidemiological data on bronchiolitis concerning viral causes and the associated clinical severity.

The investigators want to conduct a prospective cohort study, comparing incidence of co-infection and clinical severity, in two cohort: one with isolation of RS positive bronchiolitis as a separate cohort within bronchiolitis and one without isolation (all children with RS-negative bronchiolitis are nursed together independent of viral agent)

DETAILED DESCRIPTION:
Acute bronchiolitis is a major cause for hospitalisation in young children during the winter season. Human Respiratory Syncytial Virus (RSV) is the most frequently identified virus, however with the use of new and highly sensitive molecular amplification methods, the role of other viral pathogens in bronchiolitis has been increasingly recognized. Various disease severity has been shown for a range of respiratory viruses, and double viral infection is relatively common, occurring in about 10-30% of hospitalised patients. There is no consensus, however, on the impact of such co-infection on disease severity: Some studies showed more severe disease in co-infected children,while others did not.Most hospitals perform routine viral testing to identify and isolate RSV-infected infants, with the aim of reducing the risk of nosocomial cross-infection of other patients.However, no good evidence is available of how effective this approach is in preventing nosocomial cross-infections among admitted patients with the clinical diagnosis of bronchiolitis.

Because of limited isolation facilities, patients with bronchiolitis admitted to our pediatric ward initially share a room, pending the results of virological diagnosis. We hypothesize that contact isolation measures and maintaining enough distance between the beds in a shared room should be sufficient in preventing cross-infection, since the major route of transmission of respiratory viruses is by close contact with infected secretions and not by small-particle aerosol.

Objectives The purpose of this study was to determine the incidence of cross-infection in children hospitalised for bronchiolitis, when patients with RSV share the same room with patients with bronchiolitis infected with another virus during the first day of admission.

Study design The study was conducted at our 30-bed pediatric ward. From December 2011 through March 2012, all eligible infants younger than two years of age hospitalised for acute bronchiolitis were prospectively enrolled. Bronchiolitis was defined as acute respiratory disease, accompanied by coryza, cough, inspiratory crackles and/or expiratory wheezing on auscultation. Infants with chronic lung disease, congenital heart disease and Down's syndrome were excluded.

We prospectively collected the following demographic and clinical information, including presence and number of room mates, virological diagnosis of the patient and room mates, and daily dyspnoea score assessed by an independent researcher, who was unaware of virological diagnosis. A nasopharyngeal aspirate was collected for virological diagnosis by direct immunochromatographic antigen detection immediately at admission, every fourth day during admission, and five to seven days after discharge.All patients with bronchiolitis were treated with standard hygienic measures. Medical and nursing personnel wore gowns, gloves and masks during patient contact and washed their hands before and after patient contact. Parents and visitors were asked to wash hands before leaving the room. On the first day of admission, pending the results of the RSV-PCR (polymerase chain reaction), patients shared a two- or four-bed room, with beds separated at least 1,5 meter. Cohorting of RSV-infected patients commenced as soon as the result of RSV-PCR was known, generally within one day after admission.

Statistical analysis Chi-square test was used to compare categorical data, Mann-Whitney U-tests for continuous data because of skewed distributions. Statistical analyses were performed using Statistical Package for the Social Sciences (SPSS) version 19.

ELIGIBILITY:
Inclusion Criteria:

* patients under 2 years of age
* hospitalized for bronchiolitis

Exclusion Criteria:

* bronchopulmonary disease
* congenital heart defect,
* congenital pulmonary disease,
* Down's syndrome

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admittted for bronchiolitis under 2 years of age
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolita Bekhof, MD, Principal Investigator — Isala
Locations (1):
- Isala Klinieken, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 84 eligible patients, 48 were included in the study
Period: Overall Study
Arm/Group | Group Without Isolation | Group With Isolation
Started | 37 | 11
Completed | 37 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Without Isolation | Group With Isolation | Total
Number analyzed (Participants) | 37 | 11 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 11 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.4 (0.4) | 0.6 (0.5) | 0.5 (0.4)
Gender [Count of Participants; unit: Participants]
  Female | 17 | 5 | 22
  Male | 20 | 6 | 26
Region of Enrollment [Number; unit: participants]
  Netherlands | 37 | 11 | 48

OUTCOME MEASURES:

1. Primary Outcome: Duration of Hospital Stay
Time Frame: duration of hospitalisation, an average of 3-4 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group Without Isolation | Group With Isolation
Number analyzed (Participants) | 37 | 11
days | 3.9 (3.6) | 2.1 (1.2)

2. Secondary Outcome: Number of Days With Tube Feeding
Description: number of days the patient has been tube fed
Time Frame: duration of hospitalisation, an average of 3-4 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group Without Isolation | Group With Isolation
Number analyzed (Participants) | 37 | 11
days | 2.2 (3.5) | 0.7 (1.3)

3. Secondary Outcome: Supplemental Oxygen Needed
Description: number of days that supplemental oxygen was needed
Time Frame: duration of hospitalisation, an average of 3-4 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group Without Isolation | Group With Isolation
Number analyzed (Participants) | 37 | 11
days | 2.1 (2.6) | 1.1 (1.6)

4. Secondary Outcome: Highest Dyspnoea Score
Description: highest dyspnoea score (0-10) recorded during admission (0 is no dsypnoea, 10 is highest dyspnoeascore, thus the worst)
Time Frame: duration of hospitalisation, an average of 3-4 days
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | Group Without Isolation | Group With Isolation
Number analyzed (Participants) | 37 | 11
units on a scale (0-10) | 3.4 (2.1) | 2.9 (1.7)

5. Secondary Outcome: Mechanical Ventilation
Description: Mechanical ventilation and endotracheal intubation needed
Time Frame: duration of hospitalisation, an average of 3-4 days
Measure: Number; unit: participants
Arm/Group | Group Without Isolation | Group With Isolation
Number analyzed (Participants) | 37 | 11
participants | 2 | 1

6. Secondary Outcome: Cross-infection
Description: nosocomially acquired cross-infection
Time Frame: measured until 1 week after hospital exit
Measure: Number; unit: participants
Arm/Group | Group Without Isolation | Group With Isolation
Number analyzed (Participants) | 37 | 11
participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | Group Without Isolation | Group With Isolation
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/11
Other Adverse Events (participants affected / at risk) | 0/37 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No